CLINICAL TRIAL: NCT02107963
Title: A Phase I Trial of T Cells Expressing an Anti-GD2 Chimeric Antigen Receptor in Children and Young Adults With GD2+ Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 140059; 14-C-0059
Record Dates: First submitted 2014-04-05; First posted 2014-04-09 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Sarcoma; Osteosarcoma; Neuroblastoma; Melanoma
Keywords: GD2-Expressing Tumors; Anti-GD2 Chimeric Antigen Receptor; Osteosarcoma; Adoptive Immunotherapy; Sarcomas
MeSH Terms: conditions — Sarcoma; Osteosarcoma; Neuroblastoma; Melanoma | interventions — AP 1903 reagent; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Dose escalation of anti-GD2 CAR T cells
  Interventions: Biological: Anti-GD2-CAR engineered T cells; Drug: AP1903; Drug: Cyclophosphamide
- Arm 2 (Experimental): Dose expansion of anti-GD2 CAR T cells
  Interventions: Biological: Anti-GD2-CAR engineered T cells; Drug: AP1903; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: Anti-GD2-CAR engineered T cells — Administer anti-GD2 CAR T cells 1 x 105 transduced T cells/kg; 1 x 106 transduced T cells/kg; 3 x 106 transduced T cells/kg; and 1 x 107 transduced T cells/kg
Drug: AP1903 — If unacceptable toxicity occurs that is possibly, probably or likely related to anti-GD2-CAR T cells, AP1903, a dimerizing agent, may be administered to mediate clearance of the genetically engineered cells and resolve toxicity
Drug: Cyclophosphamide — 1800mg/m2/d X 2 days as a lymphodepleting regimen

SUMMARY:
Background

GD2 is a well-characterized tumor antigen in neuroblastoma, which is also expressed on osteosarcomas and some other sarcomas. T cells expressing 1st generation anti-GD2 chimeric antigen receptors (CARs) were safe and mediated modest antitumor activity in some patients with refractory neuroblastoma.

A 3rd generation anti-GD2-CAR (GD2-CAR.OX40.28.z.ICD9) has been produced and holds promise for increased activity compared to the 1st generation GD2-CAR already studied in clinical trials. As an added safety measure, the vector includes a suicide switch comprising a caspase dimerization domain (ICD9) that can be activated by a small molecule to induce death of the genetically engineered cells if they were induce untoward toxicity.

Objectives

Primary:Determine the feasibility of producing anti GD2-CAR cells meeting the established release criteria and to assess the safety of administering escalating doses of anti-GD2-CAR engineered T cells in children and young adults with GD2+ solid tumors, including neuroblastoma, following cyclophosphamide-based lymphodepletion.

Secondary:

1. Determine if administration anti-GD2-CAR engineered T cells mediate antitumor effects in children and young adults with GD2+ solid tumors;
2. Measure persistence of adoptively transferred anti-GD2-CAR T cells and correlate this with antitumor effects;
3. Extend information regarding the prevalence and intensity of GD2 expression in non-neuroblastoma, non-osteosarcoma solid tumors in children and young adults;
4. If unacceptable toxicity occurs that is possibly, probably or likely related to anti-GD2-CAR T cells, assess the capacity for AP1903, a dimerizing agent, to mediate clearance of the genetically engineered cells and resolve toxicity; and
5. Assess toxicity of AP1903 if administered to mediate clearance of anti-GD2-CAR T cells.

Eligibility

Patients 1-35 years of age, at least 15 kg, with osteosarcoma or a GD2+ solid tumor (including neuroblastoma) that has recurred after or not responded to standard therapy and is deemed incurable by standard therapy.

Design

After apheresis to collect T cells for transduction, patients receive cyclophosphamide 1800mg/m(2)/d as a lymphodepleting regimen. A phase I cell dose escalation scheme will used at 4 dose levels (1 x 10(5) transduced T cells/kg; 1 x 10(6) transduced T cells/kg; 3 x 10(6) transduced T cells/kg; and 1 x 10(7) transduced T cells/kg), using a standard 3 plus 3 dose escalation design. An expanded group of a total of 12 patients will be treated at the highest dose, comprising at least 6 osteosarcoma patients.

Patients will be monitored for toxicity, antitumor effects and persistence of anti-GD2-CAR T cells.

Patients with a PR, SD may receive a 2nd cycle at the next higher dose level a minimum of 60 days following completion of the first cycle if eligibility criteria are met.

A maximum of 36 patients may be treated on this study. Given that there is likelihood that some patients with non-osteosarcoma will not meet the criteria for GD2 expression to be eligible for enrollment, up to 72 subjects will be screened to enroll a maximum of 36 patients for treatment. Up to 2-3 patients will be accrued per month, and therefore this study may require up to 2-3 years to complete enrollment and treatment.

DETAILED DESCRIPTION:
Background

GD2 is a well-characterized tumor antigen in neuroblastoma, which is also expressed on osteosarcomas and some other sarcomas. T cells expressing 1st generation anti-GD2 chimeric antigen receptors (CARs) were safe and mediated modest antitumor activity in some patients with refractory neuroblastoma.

A 3rd generation anti-GD2-CAR (GD2-CAR.OX40.28.z.ICD9) has been produced and holds promise for increased activity compared to the 1st generation GD2-CAR already studied in clinical trials. As an added safety measure, the vector includes a suicide switch comprising a caspase dimerization domain (ICD9) that can be activated by a small molecule to induce death of the genetically engineered cells if they were induce untoward toxicity.

Objectives

* Primary:Determine the feasibility of producing anti GD2-CAR cells meeting the established release criteria and to assess the safety of administering escalating doses of anti-GD2-CAR engineered T cells in children and young adults with GD2+ solid tumors, including neuroblastoma, following cyclophosphamide-based lymphodepletion.
* Seconday: 1) Determine if administration of anti-GD2-CAR engineered T cells mediate antitumor effects in children and young adults with GD2+ solid tumors; 2) Measure persistence of adoptively transferred anti-GD2-CAR T cells and correlate this with antitumor effects; 3) Extend information regarding the prevalence and intensity of GD2 expression in non-neuroblastoma, non- osteosarcoma solid tumors in children and young adults; 4) If unacceptable toxicity occurs that is possibly, probably or likely related to anti-GD2-CAR T cells, assess the capacity for AP1903, a dimerizing agent, to mediate clearance of the genetically engineered cells and resolve toxicity; and 5) Assess toxicity of AP1903 if administered to mediate clearance of anti-GD2-CAR T cells.

Eligibility

Patients 1-35 years of age, at least 15 kg, with osteosarcoma or a GD2+ solid tumor (including neuroblastoma) that has recurred after or not responded to standard therapy and is deemed incurable by standard therapy.

Design

After apheresis to collect T cells for transduction, patients receive cyclophosphamide 1800mg/m(2)/d as a lymphodepleting regimen. A phase I cell dose escalation scheme will used at 4 dose levels (1 x 10(5) transduced T cells/kg; 1 x 10(6) transduced T cells/kg; 3 x 10(6) transduced T cells/kg; and 1 x 10(7) transduced T cells/kg), using a standard 3 plus 3 dose escalation design. An expanded group of a total of 12 patients will be treated at the highest dose, comprising at least 6 osteosarcoma patients.

Patients will be monitored for toxicity, antitumor effects and persistence of anti-GD2-CAR T cells.

Patients with a PR, SD may receive a 2nd cycle at the next higher dose level a minimum of 60 days following completion of the first cycle if eligibility criteria are met.

A maximum of 36 patients may be treated on this study. Given that there is likelihood that some patients with non-osteosarcoma will not meet the criteria for GD2 expression to be eligible for enrollment, up to 72 subjects will be screened to enroll a maximum of 36 patients for treatment. Up to 2-3 patients will be accrued per month, and therefore this study may require up to 2-3 years to complete enrollment and treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis

     (a) Osteosarcoma, neuroblastoma and melanoma that have been treated with standard frontline therapy and are judged to be incurable with standard therapy, based upon the fact that they are unresectable, metastatic, progressive/persistent or recurrent.

     Evaluable disease must be present.

     i) For all histologies except osteosarcoma and neuroblastoma, pathologic review of frozen tissue must document GD2+ expression. Positive expression is defined as at least 2+ expression (0-4+ scale) in >50 percent of the tumor cells using anti-GD2 mAb 14G2a. If adequate archived frozen tissue is available, this may be utilized, or if not, patients may undergo biopsy following enrollment to obtain tissue to assess GD2 expression, with the following restrictions.

     ii) Patients with histologies other than osteosarcoma or neuroblastoma must have adequate accessible tumor for biopsy (at least 1 cm diameter).

     iii) Procedures employed to acquire biopsies for tumor lysates will be limited to percutaneous needle or core biopsies, thoracoscopic excision or open biopsies of readily accessible lesions. Pulmonary lesions may be biopsied but extensive surgery such as thoracotomy or laparotomy should not be employed.

     iv) Patients who will require biopsy should not be enrolled if in the opinion of the principal investigator, the tumor site places the patient at substantial risk from the biopsy procedure.
  2. Weight greater than or equal to 15 kg
  3. Age less than or equal to 35 years old at the time of enrollment.
  4. Prior Therapy:

     1. The patient s malignancy must have relapsed after or failed to respond to frontline curative therapy and/or there must not be any curative treatment options available at the time of study entry.
     2. There is no limit to the number of prior treatment regimens. However, patients must have fully recovered from the acute toxic effects of prior chemotherapy, immunotherapy, or radiotherapy prior to study enrollment. Any grade 3 or 4 non-hematologic toxicity of any previous therapy must have resolved to grade 2 or less.
     3. Myelosuppressive chemotherapy: Patients must not have received myelosuppressive chemotherapy within 3 weeks of enrollment (6 weeks if prior nitrosourea).
     4. Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with a growth factor. At least 14 days must have elapsed after receiving pegfilgrastim.
     5. At least 7 days must have elapsed since the completion of therapy with a biologic agent, targeted agent, tyrosine kinease inhibitor or a metronomic nonmyelosuppressive regimen.
     6. Monoclonal antibodies: At least 4 weeks must have elapsed since prior therapy that included a monoclonal antibody.
     7. Radiotherapy: 3 weeks must have elapsed since XRT
  5. Performance status:

     ECOG 0, 1 or 2, or for children less than or equal to 10 years of age, Lansky greater than or equal to 60.
  6. Cardiac function:

     Left ventricular ejection fraction greater than or equal to 40 percent or fractional shortening greater than or equal to 28 percent.
  7. Liver function:

     Serum total bilirubin < 2 mg/dl, serum AST and ALT less than or equal to 3 x upper limit of normal. Patients with Gilbert s syndrome are excluded from the requirement of a normal bilirubin and patients will not be excluded if liver enzyme elevation is due to tumor involvement. (Gilbert s syndrome is found in 3-10% of the general population, and is characterized by mild, chronic unconjugated hyperbilirubinemia in the absence of liver disease or overt hemolysis). NOTE: Adult values will be used for calculating hepatic toxicity and determining eligibility, as is standard on POB phase I trials.
  8. Renal function:

     Age-adjusted normal serum creatinine according to the following table or a creatinine clearance greater than or equal to 60 ml/min/1.73 m(2).

     Age less than or equal to 5 Maximum serum creatinine (mg/dl) 0.8

     Age greater than 5 and less than or equal to 10 Maximum serum creatinine (mg/dl) 1.0

     Age greater than 10 and less than or equal to 15 Maximum serum creatinine (mg/dl) 1.2

     Age greater than 15 Maximum serum creatinine (mg/dl) 1.5
  9. Marrow function:

     ANC must be > 750/mm(3), platelet count must be greater than or equal to 75,000/mm(3) (not achieved by transfusion).
  10. Ability to give informed consent.

      For patients <18 years of age, their legal guardian must give informed consent. Pediatric patients will be included in age-appropriate discussion in order to obtain verbal assent.
  11. Durable power of attorney form offered (patients (Bullet)18 years of age only).
  12. Birth Control

Female and male patients (and when relevant their partners) must be willing to practice birth control (including abstinence) during and for two months after treatment, if of childbearing potential.

EXCLUSION CRITERIA:

1. Concurrent Illnesses

   Clinically significant systemic illness (e.g. serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the judgment of the PI would compromise the patient s ability to tolerate protocol therapy or significantly increase the risk of complications.

   Peripheral nerve symptoms from prior therapies or from tumor compression > grade 1.
2. Untreated CNS metastasis

   Extradural masses that have not invaded the brain parenchyma or parameningeal tumors without evidence for leptomeningeal spread will not render the patient ineligible. Patients with previous CNS tumor involvement that has been treated and is stable for at least 6 weeks following completion of therapy are eligible.
3. Prior Therapy

   Previous treatment with genetically engineered GD2-CAR T cells. Previous vaccine therapy, anti-GD2 mAb therapy or therapy with other genetically engineered T cells is not an exclusion criteria.
4. Lactating or pregnant females (due to risk to fetus or newborn).
5. Active HIV, HBV or HCV infection.
6. Immune Therapies

Patients who require systemic corticosteroid or other immunosuppressive therapy. Immunosuppressive therapy must be stopped at least 14 days prior to cell infusion.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 1 Year to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2016-08-15 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility | 29 days
  Determine the feasibility of producing anti-GD2-CAR cells meeting the established release criteria and to assess the safety of administering escalating doses of autologous anti-GD2-CAR (anti-GD2.28.z.OX40.ICD9) engineered T cells in children and young adults with osteosarcoma and GD2+ solid tumors (excluding neuroblastoma) following cyclophosphamide based lymphodepletion.

SECONDARY OUTCOMES:
Determine antitumr effects | 60 days
  Determine antitumr effects
Persistence of anti-GD2 CAR T cells and correlate with anti-tumor effects | 60 days
  Persistence of anti-GD2 CAR T cells and correlate with anti-tumor effects
Evaluate prevalence of GD2 expression | 3 years
  Evaluate prevalence of GD2 expression
Evaluate effectiveness of AP1903 to mediate clearance of anti-GD2 CAR T cells | When needed
  Evaluate effectiveness of AP1903 to mediate clearance of anti-GD2 CAR T cells
Safety | time of treatment
  Assess toxicity of AP1903

CONTACTS AND LOCATIONS:
Overall Officials: Rosandra N Kaplan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Background] Yu AL, Gilman AL, Ozkaynak MF, London WB, Kreissman SG, Chen HX, Smith M, Anderson B, Villablanca JG, Matthay KK, Shimada H, Grupp SA, Seeger R, Reynolds CP, Buxton A, Reisfeld RA, Gillies SD, Cohn SL, Maris JM, Sondel PM; Children's Oncology Group. Anti-GD2 antibody with GM-CSF, interleukin-2, and isotretinoin for neuroblastoma. N Engl J Med. 2010 Sep 30;363(14):1324-34. doi: 10.1056/NEJMoa0911123. PMID 20879881
- [Background] Lee DW, Barrett DM, Mackall C, Orentas R, Grupp SA. The future is now: chimeric antigen receptors as new targeted therapies for childhood cancer. Clin Cancer Res. 2012 May 15;18(10):2780-90. doi: 10.1158/1078-0432.CCR-11-1920. PMID 22589486
- [Background] Di Stasi A, Tey SK, Dotti G, Fujita Y, Kennedy-Nasser A, Martinez C, Straathof K, Liu E, Durett AG, Grilley B, Liu H, Cruz CR, Savoldo B, Gee AP, Schindler J, Krance RA, Heslop HE, Spencer DM, Rooney CM, Brenner MK. Inducible apoptosis as a safety switch for adoptive cell therapy. N Engl J Med. 2011 Nov 3;365(18):1673-83. doi: 10.1056/NEJMoa1106152. PMID 22047558
- [Derived] Kaczanowska S, Murty T, Alimadadi A, Contreras CF, Duault C, Subrahmanyam PB, Reynolds W, Gutierrez NA, Baskar R, Wu CJ, Michor F, Altreuter J, Liu Y, Jhaveri A, Duong V, Anbunathan H, Ong C, Zhang H, Moravec R, Yu J, Biswas R, Van Nostrand S, Lindsay J, Pichavant M, Sotillo E, Bernstein D, Carbonell A, Derdak J, Klicka-Skeels J, Segal JE, Dombi E, Harmon SA, Turkbey B, Sahaf B, Bendall S, Maecker H, Highfill SL, Stroncek D, Glod J, Merchant M, Hedrick CC, Mackall CL, Ramakrishna S, Kaplan RN. Immune determinants of CAR-T cell expansion in solid tumor patients receiving GD2 CAR-T cell therapy. Cancer Cell. 2024 Jan 8;42(1):35-51.e8. doi: 10.1016/j.ccell.2023.11.011. Epub 2023 Dec 21. PMID 38134936
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-C-0059.html